CLINICAL TRIAL: NCT00318643
Title: A Phase 1-2a, Multicenter, Open-Label, Multiple Dose, Safety, Tolerability, and Pharmacokinetic Study of Recombinant Human Hyaluronidase (Chemophase®) in Combination With Mitomycin in Patients With Non-Muscular-Invasive Bladder Cancer
Brief Title: Safety Study of Recombinant Human Hyaluronidase (Chemophase) in Combination With Mitomycin in Participants With Superficial Bladder Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Halozyme Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: HZ2-05-01
Record Dates: First submitted 2006-04-25; First posted 2006-04-27 (Estimated); Results first posted 2021-10-29 (Actual); Last update posted 2021-10-29 (Actual); Status verified 2021-09

CONDITIONS: Bladder Cancer
Keywords: Non-invasive bladder cancer; Chemophase; Intravesical administration; Superficial Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms; Non-Muscle Invasive Bladder Neoplasms | interventions — Mitomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Cohort 1: MMC plus Chemophase 20,000 U (Experimental): Participants will receive 40 milligrams (mg) MMC intravesically on Day 1 of Week 1 followed by a combination of 40 mg MMC and 20,000 U Chemophase intravesically once weekly from Weeks 2 through 6.
  Interventions: Drug: Mitomycin C; Drug: Chemophase
- Cohort 2: MMC plus Chemophase 60,000 U (Experimental): Participants will receive 40 mg MMC intravesically on Day 1 of Week 1 followed by a combination of 40 mg MMC and 60,000 U Chemophase intravesically once weekly from Weeks 2 through 6.
  Interventions: Drug: Mitomycin C; Drug: Chemophase
- Cohort 3: MMC plus Chemophase 200,000 U (Experimental): Participants will receive 40 mg MMC intravesically on Day 1 of Week 1 followed by a combination of 40 mg MMC and 200,000 U Chemophase intravesically once weekly from Weeks 2 through 6.
  Interventions: Drug: Mitomycin C; Drug: Chemophase
- Cohort 4: MMC plus Chemophase 400,000 U (Experimental): Participants will receive 40 mg MMC intravesically on Day 1 of Week 1 followed by a combination of 40 mg MMC and 400,000 U Chemophase intravesically once weekly from Weeks 2 through 6.
  Interventions: Drug: Mitomycin C; Drug: Chemophase
- Cohort 5: MMC plus Chemophase 800,000 U (Experimental): Participants will receive 40 mg MMC intravesically on Day 1 of Week 1 followed by a combination of 40 mg MMC and 800,000 U Chemophase intravesically once weekly from Weeks 2 through 6.
  Interventions: Drug: Mitomycin C; Drug: Chemophase

INTERVENTIONS:
Drug: Mitomycin C — intravesical administration
Drug: Chemophase — intravesical administration

SUMMARY:
The purpose of this study is to explore a treatment that potentially enhances the delivery of chemotherapy to tumors in participants with superficial bladder cancer. The investigational medication to be studied is an enzyme called ChemophaseTM (recombinant human hyaluronidase, rHuPH20). Chemophase is being specifically developed for use with other anticancer drug to increase the local penetration of the anticancer drug for the treatment of superficial bladder cancer. In this study, Chemophase will be given in combination with mitomycin C directly into the bladder. Mitomycin C is an anti-tumor drug that is commonly used to treat superficial bladder cancer. It is envisioned that Chemophase with mitomycin C may potentially increase the local penetration of mitomycin C into remaining cancer cells following surgery to treat superficial bladder cancer.

DETAILED DESCRIPTION:
The primary objectives of this study are to:

1. determine the maximum tolerated dose (MTD) and dose-limiting toxicities (DLTs) of escalating doses of Chemophase in combination with mitomycin (mitomycin C, MMC) administered as weekly intravesical instillations for five weeks, and
2. establish the dose of Chemophase with MMC recommended for future studies.

The secondary objectives of this study are to:

1. assess the pharmacokinetics of intravesical administration of MMC alone and in combination with intravesical administration of Chemophase,
2. for those participants treated at the MTD, assess the safety and tolerability of intravesical administration of MMC with Chemophase over up to 7 additional maintenance treatments every 3 months following the initial six weekly instillations, and
3. observe participants for any preliminary evidence of anti-tumor activity of MMC and Chemophase when combined.

Study participants will receive six weekly study treatments administered intravesically (at Weeks 1 through 6) followed by post-treatment evaluations, at Weeks 8 and 12. The 12 participants treated at MTD will continue to receive combination therapy every three months until the end of Year 2 or until the time of documented tumor recurrence, whichever occurs first. For other participants, long-term follow-up after Week 12 will consist of disease monitoring of participants by telephone and will be performed every three months beginning three months after last study treatment for two years and then every six months thereafter, until bladder tumor recurrence.

ELIGIBILITY:
Inclusion Criteria:

* Participants with initial presentation or recurrence of Stage Ta, T1 or Tis, any grade, bladder cancer after transurethral resection of bladder tumor (TURBT).
* TURBT within 42 days prior to Day 1/Week 1
* Karnofsky Performance Status greater than or equal to 80%
* Life expectancy at least 3 years
* 18 years or older
* A negative pregnancy test (if female of child-bearing potential)
* Acceptable liver function within 7 days defined as: bilirubin less than or equal to 1.5 times upper limit of normal, and aspartate aminotransferase (AST) Glutamic-oxalacetic transaminase (SGOT), alanine aminotransferase (ALT), glutamic-pyruvic transaminase (SGPT), and alkaline phosphatase <= 2.5 times upper limit of normal
* Acceptable renal function within 7 days defined as: serum creatinine less than or equal to 1.5 times upper limit of normal, or calculated creatinine clearance greater than or equal to 40 milliliter (mL)/minute/1.73 meter^2
* Acceptable hematologic status within 7 days defined as: absolute neutrophil count (ANC) greater than or equal to 2,500 cells/millimeter^3, platelet count greater than or equal to 150,000/millileter^3, and hemoglobin greater than or equal to 10.0 grams/deciliter.
* Urinalysis showing no clinically significant abnormalities except those attributable to bladder cancer.
* For men and women of child-producing potential, agreement to use an effective contraceptive method during the treatment period of the study.
* Signed, written Institutional Review Board (IRB)-approved informed consent

Exclusion Criteria:

* History or previous diagnosis of bladder fibrosis
* Total bladder capacity estimated at cystoscopy to be less than 150 mL
* Urinary incontinence of a severity that would compromise the ability of the participant to retain the study drug intravesical instillation for two hours.
* Severe irritative voiding symptoms such as urgency, frequency, or nocturia
* Known other malignant disease except squamous or basal cell skin cancer unless the malignancy has been in complete remission off therapy for at least 5 years.
* Major surgery, other than TURBT and diagnostic surgery, within 28 days prior to Day 1/Week 1.
* Active, uncontrolled bacterial, viral, or fungal infections, including urinary tract infection.
* Treatment with radiation therapy, surgery, chemotherapy, or investigational therapy within one month prior to Day 1/Week 1 on study (two months for nitrosureas or MMC), unless given as standard treatment for bladder cancer and provided that patient is free of all treatment-related toxicities as of Day 1/Week 1.
* Known infection with human immunodeficiency virus (HIV)
* Known active infection with hepatitis B or hepatitis C
* Serious disease (e.g., hydronephrosis, liver failure, or other conditions) that could compromise protocol objectives in the opinion of the Investigator and/or the Sponsor (Halozyme).
* History of a hypersensitivity or idiosyncratic reaction to, or other contraindication to, mitomycin.
* Known allergy to bee or vespid venom
* Known coagulation disorder or bleeding tendency
* Treatment with heparin or anticipation of heparin treatment during the treatment period in this study.
* Unwillingness or inability to comply with procedures required in this protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2006-03-30 (Actual); Primary Completion 2009-08-11 (Actual); Study Completion 2009-08-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - BCG Oncology, Phoenix, Arizona
  - MedResearch, La Mesa, California
  - Malcolm Randall Veterans Administration Urology Section (112-C), Gainesville, Florida
  - Advanced Research Institute, New Port Richey, Florida
  - James A. Haley Veterans Hospital, Tampa, Florida

REFERENCES:
- See also: Sponsor's website — http://www.halozyme.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1: MMC Plus Chemophase 20,000 U: Participants received 40 milligrams (mg) mitomycin C (MMC) intravesically on Day 1 of Week 1 followed by a combination of 40 mg MMC and 20,000 Units (U) Chemophase intravesically once weekly from Weeks 2 through 6.
- Cohort 2: MMC Plus Chemophase 60,000 U: Participants received 40 mg MMC intravesically on Day 1 of Week 1 followed by a combination of 40 mg MMC and 60,000 U Chemophase intravesically once weekly from Weeks 2 through 6.
- Cohort 3: MMC Plus Chemophase 200,000 U: Participants received 40 mg MMC intravesically on Day 1 of Week 1 followed by a combination of 40 mg MMC and 200,000 U Chemophase intravesically once weekly from Weeks 2 through 6.
- Cohort 4: MMC Plus Chemophase 400,000 U: Participants received 40 mg MMC intravesically on Day 1 of Week 1 followed by a combination of 40 mg MMC and 400,000 U Chemophase intravesically once weekly from Weeks 2 through 6.
- Cohort 5: MMC Plus Chemophase 800,000 U: Participants received 40 mg MMC intravesically on Day 1 of Week 1 followed by a combination of 40 mg MMC and 800,000 U Chemophase intravesically once weekly from Weeks 2 through 6.
Period: Overall Study
Arm/Group | Cohort 1: MMC Plus Chemophase 20,000 U | Cohort 2: MMC Plus Chemophase 60,000 U | Cohort 3: MMC Plus Chemophase 200,000 U | Cohort 4: MMC Plus Chemophase 400,000 U | Cohort 5: MMC Plus Chemophase 800,000 U
Started | 3 | 3 | 6 | 3 | 12
Received at Least 1 Dose of Study Drug | 3 | 3 | 6 | 3 | 12
Completed | 3 | 3 | 6 | 3 | 9
Not Completed | 0 | 0 | 0 | 0 | 3
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1
Not completed — Participant's Decision | 0 | 0 | 0 | 0 | 1
Not completed — Investigator's Decision | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Cohort 1: MMC Plus Chemophase 20,000 U: Participants received 40 mg MMC intravesically on Day 1 of Week 1 followed by a combination of 40 mg MMC and 20,000 U Chemophase intravesically once weekly from Weeks 2 through 6.
- Total: Total of all reporting groups
Arm/Group | Cohort 1: MMC Plus Chemophase 20,000 U | Cohort 2: MMC Plus Chemophase 60,000 U | Cohort 3: MMC Plus Chemophase 200,000 U | Cohort 4: MMC Plus Chemophase 400,000 U | Cohort 5: MMC Plus Chemophase 800,000 U | Total
Number analyzed (Participants) | 3 | 3 | 6 | 3 | 12 | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.7 (11.24) | 67.0 (8.54) | 65.7 (10.33) | 73.7 (3.79) | 68.0 (10.54) | 67.9 (9.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 2 | 0 | 3 | 7
  Male | 3 | 1 | 4 | 3 | 9 | 20

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) of Chemophase in Combination With MMC
Description: The MTD was defined as the maximum dose level at which no more than two of six participants experienced dose-limiting toxicities (DLT). DLT was defined as any of the following:
  * Plasma MMC concentration greater than or equal to (>=) 100 nanograms (ng)/milliliter (mL)
  * Adverse event (AE) with a Common Toxicity Criteria (CTC) grade greater than or equal to 3
  * New, treatment-emergent diagnosis of bladder fibrosis.
Time Frame: 5 weeks (Week 2 to Week 6)
Population: The Intent-To-Treat (ITT) Set included all participants who received one or more doses of Chemophase with MMC.
Measure: Number; unit: Units
Arm/Group | Cohort 5: MMC Plus Chemophase 800,000 U
Number analyzed (Participants) | 12
Units | 800000

2. Primary Outcome: Number of Participants With Dose Limiting Toxicities (DLTs)
Description: DLT was defined as any of the following:
  * Plasma MMC concentration >= 100 ng/mL
  * AE with a CTC grade greater than or equal to 3
  * New, treatment-emergent diagnosis of bladder fibrosis.
Time Frame: 5 weeks (Week 2 to Week 6)
Population: ITT Set included all participants who received one or more doses of Chemophase with MMC.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: MMC Plus Chemophase 20,000 U | Cohort 2: MMC Plus Chemophase 60,000 U | Cohort 3: MMC Plus Chemophase 200,000 U | Cohort 4: MMC Plus Chemophase 400,000 U | Cohort 5: MMC Plus Chemophase 800,000 U
Number analyzed (Participants) | 3 | 3 | 6 | 3 | 12
Participants | 0 | 0 | 1 | 0 | 0

3. Primary Outcome: Recommended Dose of Chemophase With MMC For Future Studies
Time Frame: 5 weeks (Week 2 to Week 6)
Population: ITT Set included all participants who received one or more doses of Chemophase with MMC.
Measure: Number; unit: Units
Arm/Group | Cohort 5: MMC Plus Chemophase 800,000 U
Number analyzed (Participants) | 12
Units | 800000

4. Secondary Outcome: Number of Participants With a Quantifiable MMC Plasma Concentration Value
Description: A quantifiable MMC plasma concentration value was a value that was not below the quantifiable limit (BQL) of <10.0 nanogram/milliliter (ng/mL).
Time Frame: 0 (predose), 1, 2, and 3 hours postdose at Weeks 1, 2, 5, and 6
Population: ITT Set included all participants who received one or more doses of Chemophase with MMC.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: MMC Plus Chemophase 20,000 U | Cohort 2: MMC Plus Chemophase 60,000 U | Cohort 3: MMC Plus Chemophase 200,000 U | Cohort 4: MMC Plus Chemophase 400,000 U | Cohort 5: MMC Plus Chemophase 800,000 U
Number analyzed (Participants) | 3 | 3 | 6 | 3 | 12
Participants
  Week 1: Predose | 0 | 0 | 0 | 0 | 0
  Week 1: 1 hour | 0 | 0 | 0 | 0 | 1
  Week 1: 2 hours | 0 | 0 | 0 | 0 | 1
  Week 1: 3 hours | 0 | 0 | 0 | 0 | 0
  Week 2: Predose | 0 | 0 | 0 | 0 | 0
  Week 2: 1 hour | 0 | 0 | 0 | 0 | 0
  Week 2: 2 hours | 0 | 0 | 0 | 0 | 0
  Week 2: 3 hours | 0 | 0 | 0 | 0 | 0
  Week 5: Predose | 0 | 0 | 0 | 0 | 0
  Week 5: 1 hour | 0 | 0 | 0 | 0 | 0
  Week 5: 2 hours | 0 | 0 | 1 | 0 | 0
  Week 5: 3 hours | 0 | 0 | 1 | 0 | 0
  Week 6: Predose | 0 | 0 | 0 | 0 | 0
  Week 6: 1 hour | 0 | 0 | 0 | 1 | 0
  Week 6: 2 hours | 0 | 0 | 0 | 1 | 0
  Week 6: 3 hours | 0 | 0 | 0 | 0 | 0

5. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Description: TEAEs were defined as any AE that occurred after the first administration of the study drug and until the end of the study. AEs were defined as any untoward medical occurrence in a participant administered study drug and that did not necessarily have a causal relationship with the study drug. SAEs were defined as any AE that, in the view of either the Investigator or Sponsor, resulted in any of the following outcomes as fatal, life-threatening, required in-participant hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, a congenital anomaly/birth defect, an important medical event. A summary of all SAEs and Other AEs (nonserious) regardless of causality is located in 'Reported Adverse Events' Section.
Time Frame: Baseline up to 2 years
Population: The Safety Set included all participants who received one or more doses of Chemophase.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: MMC Plus Chemophase 20,000 U | Cohort 2: MMC Plus Chemophase 60,000 U | Cohort 3: MMC Plus Chemophase 200,000 U | Cohort 4: MMC Plus Chemophase 400,000 U | Cohort 5: MMC Plus Chemophase 800,000 U
Number analyzed (Participants) | 3 | 3 | 6 | 3 | 12
Participants
  TEAEs | 1 | 1 | 4 | 2 | 10
  SAEs | 1 | 0 | 2 | 0 | 2

6. Secondary Outcome: Number of Participants Who Remained Tumor Free at the End of the Study
Time Frame: Baseline up to 2 years
Population: ITT Set included all participants who received one or more doses of Chemophase with MMC.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: MMC Plus Chemophase 20,000 U | Cohort 2: MMC Plus Chemophase 60,000 U | Cohort 3: MMC Plus Chemophase 200,000 U | Cohort 4: MMC Plus Chemophase 400,000 U | Cohort 5: MMC Plus Chemophase 800,000 U
Number analyzed (Participants) | 3 | 3 | 6 | 3 | 12
Participants | 2 | 0 | 2 | 1 | 6

ADVERSE EVENTS:
Time Frame: Baseline up to 2 years
Description: The Safety Set included all participants who received one or more doses of Chemophase.
Arm/Group | Cohort 1: MMC Plus Chemophase 20,000 U | Cohort 2: MMC Plus Chemophase 60,000 U | Cohort 3: MMC Plus Chemophase 200,000 U | Cohort 4: MMC Plus Chemophase 400,000 U | Cohort 5: MMC Plus Chemophase 800,000 U
Serious Adverse Events (participants affected / at risk) | 1/3 | 0/3 | 2/6 | 0/3 | 2/12
Other Adverse Events (participants affected / at risk) | 0/3 | 1/3 | 4/6 | 2/3 | 10/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: MMC Plus Chemophase 20,000 U (N=3) | Cohort 2: MMC Plus Chemophase 60,000 U (N=3) | Cohort 3: MMC Plus Chemophase 200,000 U (N=6) | Cohort 4: MMC Plus Chemophase 400,000 U (N=3) | Cohort 5: MMC Plus Chemophase 800,000 U (N=12)
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Small cell lung cancer stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Angina unstable (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: MMC Plus Chemophase 20,000 U (N=3) | Cohort 2: MMC Plus Chemophase 60,000 U (N=3) | Cohort 3: MMC Plus Chemophase 200,000 U (N=6) | Cohort 4: MMC Plus Chemophase 400,000 U (N=3) | Cohort 5: MMC Plus Chemophase 800,000 U (N=12)
Urinary tract infection (Infections and infestations) | 0 | 1 | 2 | 0 | 2
Asymptomatic bacteriuria (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Folliculitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Helicobacter infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Onychomycosis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
Cerebral ischaemia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Diabetic retinopathy (Eye disorders) | 0 | 0 | 0 | 0 | 1
Dry eye (Eye disorders) | 0 | 0 | 0 | 0 | 1
Eye pain (Eye disorders) | 0 | 0 | 0 | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Diverticulum (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Dysuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 2
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 2
Bladder spasm (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Calculus urethral (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Micturition urgency (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Nocturia (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Urethral disorder (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Urtheral haemorrhage (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Genital rash (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 1
Balanitis (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0
Prostatitis (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 1
Malaise (General disorders) | 0 | 0 | 0 | 0 | 1
Suprapubic pain (General disorders) | 0 | 0 | 0 | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 1 | 0 | 1
Red blood cells urine positive (Investigations) | 0 | 0 | 1 | 1 | 0
White blood cells urine positive (Investigations) | 0 | 0 | 1 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 1
Blood urine present (Investigations) | 0 | 0 | 0 | 1 | 0
False positive laboratory result (Investigations) | 0 | 0 | 1 | 0 | 0
Haemoglobin decreased (Investigations) | 0 | 0 | 1 | 0 | 0
Liver function test abnormal (Investigations) | 0 | 0 | 1 | 0 | 0
White blood cells urine (Investigations) | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI must submit a copy of the proposed publication to the Sponsor 40 days prior to date of submission for publication. They can request a delay of up to 45 days if it is determined there is any patentable subject matter or confidential Information. Sponsor can make changes to the communication to remove sponsor's confidential information from it prior to publication.

DOCUMENTS (2):
  • Study Protocol (2009-02-26): https://cdn.clinicaltrials.gov/large-docs/43/NCT00318643/Prot_000.pdf
  • Statistical Analysis Plan (2008-01-11): https://cdn.clinicaltrials.gov/large-docs/43/NCT00318643/SAP_001.pdf